CLINICAL TRIAL: NCT01698502
Title: Does Physical Training Effect the Incretin Effect
Brief Title: Physical Training and the Incretin Effect
Acronym: EXINT2
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Michael Taulo Lund, MD. PhD. Student, University of Copenhagen
Other Study IDs: EXINT2_FD
Record Dates: First submitted 2012-09-26; First posted 2012-10-03 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: Incretin; Training; Glucagon like peptide; glucose dependent insulinotropic peptide; Gut; Exercise; Insulin; Focus:; Gut hormone; adaptations
MeSH Terms: conditions — Motor Activity; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Human plasma samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Trained: Healthy, Endurance trained (Maximal oxygen uptake (VO2max), ml*min-1*kg-1>60), 20-30 year, BMI: 18,5-25kg/m2, males.
- Untrained: Healthy, sedentary (Maximal oxygen uptake (VO2max), ml*min-1*kg-1<50), 20-30 year, BMI: 18,5-25kg/m2, males.

SUMMARY:
It is well known that continuous physical exercise leads to a number of changes in the body. Maximal oxygen uptake; the heart's pumping ability and muscle mass and strength increases. Also the metabolism adapts: The ability to oxidize fat increase and the insulin sensitivity in primarily in muscle, but also in the liver increase.

Also endocrine glands adapts according to the level of physical activity. It is known that in healthy, younger people the insulin secretion from the pancreas after administration of sugar consumed orally or given directly into a vein, is significantly lower in trained individuals compared with untrained. This change does, however, not only apply to glucose, as also stimulation by the amino acid arginine, shows the same pattern.

It seems plausible that the endocrine glands/cells adapts to the level of physical training, but this has not yet been investigated.

The gastrointestinal tract is the birthplace of a variety of hormones. One group of these is called incretin hormones. They stimulate the glucose dependant insulin secretion in the pancreas and affect hunger/satiety. Whether the incretin production and thus their concentration in the blood is regulated by physical training is unknown.

Obese and patients with type 2 diabetes, has, in contrast to well-trained, decreased insulin sensitivity. As a consequence their (type 2 diabetics, at least early in their disease course) meal stimulated insulin release is greater than in healthy, normal weight individuals. This in spite of the fact that the incretin effect is reduced in obese people and patients with type 2 diabetes compared to healthy, normal weight.

Whether physical training affects both the secretion of incretins and the incretin effect has not yet been studied.

The purpose of this study is to investigate whether incretin hormones in physical well-trained young men have a changed effect on insulin secretion from the pancreas compared to untrained young men. A difference may indicate that the body's endocrine glands adapts to training mode.

The investigators hypothesis is that incretin hormones have a decreased effect on the glucose dependant insulin release in physically trained persons and thus results in a lower insulin release at any given plasma glucose level.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary: 50>Maximal oxygen uptake (VO2max), ml*min-1*kg-1 OR endurance trained VO2max, ml*min-1*kg-1>60
* 20-30 years
* BMI: 18,5-25kg/m2
* Caucasian
* Healthy

Exclusion Criteria:

* Any kind of medication or diabetes in the family (parents, siblings),
* Non-caucasian

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Danish University Students from University of Copenhagen,
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Dela, Prof. MD, Study Chair — University of Copenhagen, Dep. of Biomedical Sciences, Center of healthy Ageing, XLAB
Locations (1):
- University of Copenhagen, Faculty of Health Sciences, Copenhagen, North, Denmark

REFERENCES:
- [Background] Dela F, Handberg A, Mikines KJ, Vinten J, Galbo H. GLUT 4 and insulin receptor binding and kinase activity in trained human muscle. J Physiol. 1993 Sep;469:615-24. doi: 10.1113/jphysiol.1993.sp019833. PMID 8271219
- [Background] Dela F, Mikines KJ, von Linstow M, Secher NH, Galbo H. Effect of training on insulin-mediated glucose uptake in human muscle. Am J Physiol. 1992 Dec;263(6):E1134-43. doi: 10.1152/ajpendo.2006.263.6.E1134. PMID 1476187
- [Background] Mikines KJ, Sonne B, Farrell PA, Tronier B, Galbo H. Effect of training on the dose-response relationship for insulin action in men. J Appl Physiol (1985). 1989 Feb;66(2):695-703. doi: 10.1152/jappl.1989.66.2.695. PMID 2651385
- [Background] Dela F, Mikines KJ, Von Linstow M, Galbo H. Effect of training on response to a glucose load adjusted for daily carbohydrate intake. Am J Physiol. 1991 Jan;260(1 Pt 1):E14-20. doi: 10.1152/ajpendo.1991.260.1.E14. PMID 1987787
- [Background] King DS, Dalsky GP, Staten MA, Clutter WE, Van Houten DR, Holloszy JO. Insulin action and secretion in endurance-trained and untrained humans. J Appl Physiol (1985). 1987 Dec;63(6):2247-52. doi: 10.1152/jappl.1987.63.6.2247. PMID 3325486
- [Background] Mikines KJ, Sonne B, Tronier B, Galbo H. Effects of training and detraining on dose-response relationship between glucose and insulin secretion. Am J Physiol. 1989 May;256(5 Pt 1):E588-96. doi: 10.1152/ajpendo.1989.256.5.E588. PMID 2655469
- [Background] Dupre J, Ross SA, Watson D, Brown JC. Stimulation of insulin secretion by gastric inhibitory polypeptide in man. J Clin Endocrinol Metab. 1973 Nov;37(5):826-8. doi: 10.1210/jcem-37-5-826. No abstract available. PMID 4749457
- [Background] Holst JJ, Orskov C, Nielsen OV, Schwartz TW. Truncated glucagon-like peptide I, an insulin-releasing hormone from the distal gut. FEBS Lett. 1987 Jan 26;211(2):169-74. doi: 10.1016/0014-5793(87)81430-8. PMID 3542566
- [Background] Nauck MA, Heimesaat MM, Orskov C, Holst JJ, Ebert R, Creutzfeldt W. Preserved incretin activity of glucagon-like peptide 1 [7-36 amide] but not of synthetic human gastric inhibitory polypeptide in patients with type-2 diabetes mellitus. J Clin Invest. 1993 Jan;91(1):301-7. doi: 10.1172/JCI116186. PMID 8423228
- [Background] Knop FK, Aaboe K, Vilsboll T, Volund A, Holst JJ, Krarup T, Madsbad S. Impaired incretin effect and fasting hyperglucagonaemia characterizing type 2 diabetic subjects are early signs of dysmetabolism in obesity. Diabetes Obes Metab. 2012 Jun;14(6):500-10. doi: 10.1111/j.1463-1326.2011.01549.x. Epub 2012 Jan 17. PMID 22171657

RESULTS

PARTICIPANT FLOW:
Groups:
- Trained: Healthy, Endurance trained (VO2max, ml*min-1*kg-1>60), 20-30 year, BMI: 18,5-25kg/m2, males.
- Untrained: Healthy, sedentary (VO2max, ml*min-1*kg-1<50), 20-30 year, BMI: 18,5-25kg/m2, males.
Period: Overall Study
Arm/Group | Trained | Untrained
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trained | Untrained | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (3) | 25 (3) | 25 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  Denmark | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Incretin Effect (the % of Insulin Secreted Due to the Release of the Intestinal Hormones Glucagon Like Peptide-1 (GLP-1 and Glucose-dependent Insulinotropic Peptide (GIP))
Description: The Incretin effect (the % of insulin secreted due to the release of the intestinal hormones GLP-1 and GIP) is calculated as the difference between the insulin concentration during a 3 hour oral glucose tolerance test (OGTT) (day 1) compared to a 3 hour isoglycemic intravenous glucose infusion (IIGI) (day 2) that has similar glucose excursions.
Time Frame: Test day 1 and 2 within 7 days.
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Trained | Untrained
Number analyzed (Participants) | 11 | 10
percentage | 72 (4) | 67 (3)

2. Secondary Outcome: The Total Glucose-dependent Insulinotropic Peptide (GIP) Response Measured as Area Under the GIP Curve (AUC GIP).
Description: Comparison of the total release of GIP during the 3 hour OGTT and IIGI.
Time Frame: Test day 1 and 2 within 7 days.
Measure: Mean (Standard Error); unit: pmol/L * 210 min
Arm/Group | Trained | Untrained
Number analyzed (Participants) | 11 | 10
pmol/L * 210 min
  Post OGTT | 3978 (565) | 3819 (452)
  Post IIGI | 692 (103) | 725 (202)

ADVERSE EVENTS:
Arm/Group | Trained | Untrained
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No